CLINICAL TRIAL: NCT03648320
Title: A Single Arm Phase II Efficacy Study of Peanut Oral Immunotherapy in Adults
Brief Title: The Grown Up Peanut Immunotherapy Study
Acronym: GUPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); King's College London (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 225583
Record Dates: First submitted 2018-08-06; First posted 2018-08-27 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Peanut Allergy
Keywords: IgE mediated peanut allergy; Oral immunotherapy; Desensitisation; GUPI
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peanut oral immunotherapy (Experimental): Desensitisation using peanut flour
  Interventions: Other: Peanut oral immunotherapy

INTERVENTIONS:
Other: Peanut oral immunotherapy — Daily doses of peanut flour (with 2-weekly incremental interval)

SUMMARY:
To determine efficacy and safety of peanut oral immunotherapy in adults with peanut allergy.

DETAILED DESCRIPTION:
25 adults with peanut allergy, as confirmed by double blind placebo controlled food challenge (DBPCFC), will undergo peanut oral immunotherapy (OIT) with peanut flour.

An additional 15 untreated peanut allergic adults will be recruited as comparator group for skin prick tests and mechanistic studies/immunological assays.

ELIGIBILITY:
Inclusion Criteria:

For peanut OIT patients:

Adults aged 18-40 years with:

1. A positive skin prick test to peanut extract.
2. Elevated (>0.35) serum specific Immunoglobulin E (IgE) to Ara h 2 major peanut allergen within 2 years of date of initial screening visit.
3. Positive DBPCFC to 300mg or less of peanut protein.
4. Where appropriate, use of effective form of birth control by females for the duration of participation in the study (i.e. up to exit DBPCFC).
5. Participants with asthma may be included if well controlled:

   * Asthma control questionnaire (ACQ) score <1
   * Maximum permitted asthma treatment: moderate dose of inhaled corticosteroid (ICS) and long-acting beta agonists (LABA) as treatment
   * Pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1) >80% of predicted value at screening visit
   * For asthmatic participants with intermittent mild symptoms (induced by exercise, animals or pollens) using as required salbutamol only, treatment will be given with regular low dose inhaled corticosteroids (ICS) prior to challenges and for the duration of updosing as an additional measure.

For mechanistic sub-study subjects:

Adults aged 18-40 years with:

1. A positive skin prick test to peanut extract within previous 12 months
2. Elevated serum specific IgE (>0.35) to Ara h 2 major peanut allergen within 2 years of date of initial screening visit.
3. Clinical diagnosis of peanut allergy made by an experienced allergy specialist.

Exclusion Criteria:

For peanut OIT patients:

1. Anaphylaxis to a food other than peanut - despite attempted avoidance - within the last 2 years.
2. History of life-threatening anaphylaxis or angioedema, including previous intensive care unit (ITU) admission attributable peanut allergy.
3. Asthmatic treated with higher than moderate dose of ICS (>800 mcg equivalent of beclomethasone dipropionate (BDP) per day).
4. Any asthmatic if uncontrolled or difficult to control as evidenced by any following: ACQ>1; FEV1 <80% predicted; FEV1/ forced vital capacity (FVC) <0.7 irrespective of treatment; hospital attendance (A&E or admission) for asthma in the past 2 years; treatment of asthma with oral steroids within last 2 years.
5. Evidence of non-adherence with asthma treatment from General PRactitioner (GP) repeat prescription records.
6. Participants who react to less than 1 mg of peanut protein on DBPCFC, or who cannot tolerate at least an initial dose of 1.5 mg peanut protein on OIT initiation day.
7. Participants who react to placebo during DBPCFC.
8. Ongoing treatment with beta-blockers, biologics (such as omalizumab or mepolizumab) or systemic immunosuppressive treatment.
9. Regular ongoing use of NSAIDs for a chronic condition (NSAIDs may act as a co-factor for allergic reactions)
10. For females a positive serum or urine pregnancy test with sensitivity of less than 50 mIU/mL within 72 hours of first administration of study therapy.
11. Lactating females.
12. The use of any investigational drug within 30 days of the screening visit.
13. Past history of eosinophilic oesophagitis or chronic gastro-oesophageal reflux symptoms requiring regular treatment with anti-acids.
14. Inability to discontinue antihistamines for a minimum of 4 days prior to DBPCFC visits
15. The presence of any medical condition that the investigator deems incompatible with participation in the trial.
16. Individuals with insufficient understanding of the trial.

For mechanistic sub-study subjects:

1. Ongoing treatment with biologic or systemic immunosuppressive treatment.
2. Known current pregnancy
3. Lactating females.
4. The use of any investigational drug within 30 days of the screening visit.
5. Inability to discontinue antihistamines for a minimum of 4 days prior to venesection.
6. The presence of any medical condition that the investigator deems incompatible with participation in the study.
7. Individuals with insufficient understanding of the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Desensitisation to 1.4g peanut | 7-8 months
  Tolerance of cumulative dose of 1.4g peanut protein without reaction on DBPCFC post OIT after minimum of 1 month maintenance dosing on peanut OIT

SECONDARY OUTCOMES:
Desensitisation to 4.4g peanut | 7-8 months
  Tolerance of cumulative dose of 4.4 g peanut protein without reaction on DBPCFC post OIT
Incidence of adverse events related to treatment (safety) | 7-8 months
  Incidence of local and systemic reactions during peanut OIT updosing and maintenance
Reactions with ara h 8 sensitisation | 7-8 months
  Comparison of local and systemic reactions in Ara h 8 sensitised vs. non-sensitised subjects.
Skin prick test reactivity | 9 months
  Change in size of wheal diameter to peanut extract following OIT
Immunoglobulin G (IgG) levels | 9 months
  Change in peanut-specific IgG following OIT
Quality of life measure | 7-8 months
  Change measured using Food Allergy Quality of Life Questionnaire- Adult Form (FAQLQ-AF) and the Food Allergy Independent Measure Adult Form (FAIM-AF). These are validated questionnaires consisting of 29 (FAQLQ-AF) and 6 (FAIM-AF) questions each scored on a 7 point likert scale. The total scores are the mean score of all items with a range of 1 'no impairment' to 7 'maximal impairment'.
Food Neophobia score | 7-8 months
  Change measured using validated Food Neophobia Scale (FNS) questionnaire. This consists of 8 questions with answers on a 7 point likert scale ranging from 1 ("disagree strongly") to 7 ("agree strongly"). The total score is the mean score of all questions with lower score signifying increased food neophobia.
Food Situations score | 7-8 months
  Change using Food Situations Questionnaire, validated in children and amended to be appropriate for adults. 10 different scenarios related to food are rated from 1 (very unhappy) to 5 (very happy), giving a total possible score of 50. Higher scores are indicative of lower food neophobia.
Study compliance | 7-8 months
  Compliance with OIT measured using monthly diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Till, MA FRCP PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust / King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Hunter H, Ue KL, Cornelius V, Yung CC, Thomas I, Tsilochristou O, Layhadi J, Siew LQC, Venter C, Shamji MH, Till SJ. Oral Immunotherapy in Peanut-Allergic Adults Using Real-World Materials. Allergy. 2025 Aug;80(8):2310-2318. doi: 10.1111/all.16493. Epub 2025 Apr 23. PMID 40268292